CLINICAL TRIAL: NCT06341348
Title: The Effectiveness of Case Management for Patients With Rheumatoid Arthritis in Taiwan
Brief Title: Effects of Case Management for Patients With Rheumatoid Arthritis in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Dalin Tzuchi Hospital
Record Dates: First submitted 2017-03-10; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Case Management; Rheumatoid Arthritis; Effectiveness
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Case Management

STUDY DESIGN:
Masking Description: A trained interviewer, who was blind with the study design and participants, was assigned to collect the participants' information on demographic and disease characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of case management for rheumatoid arthritis cases (Other): Case management (CM) applied is multi-component interventions, that comprised the provision of health education and professional advice, referring the client to another health care team, discussing a daily life plan, making reservations, and follow-up by telephone.
  As the control group, they received usual health education lasting for about 15 minutes per medical visit from ward nurses, which consisted of consultation in terms of disease symptoms, related treatments or the doctor's orders. They were also free to ask questions of the research team, their ward nurses and physicians at any time within the study period.
  Interventions: Other: Case management

INTERVENTIONS:
Other: Case management — Case Management (CM) is multi-component interventions, that comprised the provision of health education and professional advice, referring the client to another health care team, discussing a daily life plan, making reservations, and follow-up by telephone. All interventions were delivered by a nursing case manager who had over 5 years of nursing experience and received more than 20 hours of CM training.

SUMMARY:
Case management (CM) has been recommended as a way of inspiring measurable changes in individual behaviors and improving clinical outcomes for patients with chronic diseases. However, data on its effectiveness for Taiwanese patients with rheumatoid arthritis (RA) are limited. This study aimed to determine the long-term effectiveness of CM that focused on nurses' role among Taiwanese RA patients.

A quasi-experimental pre-post test, control-group study with purposive sampling recruited RA patients from a hospital in Taiwan during 2016-2017. CM program was composed of health education sessions and follow-up telephone consultations over a six-month period. A review of medical records and structured questionnaires yielded data about patient demographics and disease characteristics, and included Chinese version of the Arthritis Self-Efficacy Scale and the Taiwanese Depression Questionnaire. A comparison of the long-term effectiveness of the CM program was made using generalized estimating equation.

This evidence-based study may be beneficial to characterize the long-term effectiveness of CM for Taiwanese patients with RA, and may be a reference for healthcare providers in facilitating the provision of appropriate interventions to improve the adaptation processes and clinical outcomes for them.

DETAILED DESCRIPTION:
Nurse-led case management integrates a multi-component intervention comprised of health education and professional advice, as well as referral of clients to other health care team members, discussion of daily life plans, making an appointment for the next clinic, and conducting follow-up sessions by telephone.

ELIGIBILITY:
Inclusion Criteria:

* being at least 20 years old at the time of recruitment
* being able to express opinions in either Mandarin or Taiwanese, and
* having a diagnosis of rheumatoid arthritis (RA).

Exclusion Criteria:

* Those having no cognitive impairment and severe complications will be excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Time 1 (T1): prior to the CM intervention; Time 2 (T2): three days after the CM completion, and Time 3 (T3): three months after CM intervention.
  Assessed by Taiwanese Depression Questionnaire
Self-efficacy level | Time 1 (T1): prior to the CM intervention; Time 2 (T2): three days after the CM completion, and Time 3 (T3): three months after CM intervention.
  Assessed by Arthritis Self-Efficacy Scale
Sexual dysfunctionform-14 | Time 1 (T1): prior to the CM intervention; Time 2 (T2): three days after the CM completion, and Time 3 (T3): three months after CM intervention.
  Assessed by Changes in Sexual Functioning Questionnaire
DAS28 | Time 1 (T1): prior to the CM intervention; Time 2 (T2): three days after the CM completion, and Time 3 (T3): three months after CM intervention.
  Measured by Disease Activity Score of 28

IPD SHARING:
Plan to Share IPD: No